CLINICAL TRIAL: NCT04638543
Title: A Randomized, Double-Blind, Dose-Ranging, Placebo-Controlled, Multicenter, Phase 2a Study to Assess the Efficacy, Safety, and Pharmacokinetics of ABP-671 Monotherapy in Patients With Gout or Hyperuricemia
Brief Title: A Study to Assess the Efficacy, Safety, and Pharmacokinetics of ABP-671 in Patients With Gout or Hyperuricemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atom Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ABP-671-201
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Gout; Hyperuricemia
MeSH Terms: conditions — Gout; Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABP-671 (Experimental): The study will consist of three sequential groups with escalating total daily ABP-671 doses. Each group is further divided into two dose cohorts with either QD or BID dosing.
  Interventions: Drug: ABP-671
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ABP-671 — ABP-671 Tablet
  Arms: ABP-671
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a, multicenter, randomized, double-blind, placebo-controlled, dose-ranging study to evaluate the efficacy, safety, and pharmacokinetics study of 6 different dose regimens of ABP-671 compared with placebo. The study will consist of three sequential groups with escalating total daily ABP-671 doses. Each group is further divided into two dose cohorts with either QD or BID dosing. Each dose group will have 3 stages following screening: Run-in, Dose Evaluation, and Follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to understand the study procedures, the risks involved and willing to provide written informed consent before the first study related activity.
* Subject meets the diagnosis of gout as per the American College of Rheumatism/ European League Against Rheumatism (EULAR) Gout Classification Criteria or diagnosis of hyperuricemia.
* Subject has an sUA level ≥ 7.0 mg/dL at baseline.
* Subject must be willing to discontinue any other UA-lowering medication (e.g., allopurinol, febuxostat, and probenecid) and take gout prophylaxis medication during the study.
* Body mass index (BMI) ≤ 40 kg/m2.

Exclusion Criteria:

* Subject with a documented history of rheumatoid arthritis or other autoimmune disease.
* Subject with any clinically significant hepatic, cardiovascular, renal, neoplastic, psychiatric illness, or hematological disorders such as polycythemia vera, sickle cell disease, or myelodysplastic disorder.
* Subject with a history of alcohol or drug abuse within the past 1 year prior to screening, or current evidence of substance dependence or abuse.
* Subject with a positive test for active hepatitis B, hepatitis C infection or human immunodeficiency virus (HIV) infection.
* Subject with active liver disease, or hepatic dysfunction.
* Subject with an inadequate renal function with estimated serum creatinine > 1.5 mg/dL (> 0.133 mmol/L) or creatinine clearance < 60 mL/min (by Cockcroft-Gault formula).
* Subject with a history of malignancy within the previous 5 years with the exception of non-melanoma skin cancer that has been treated with no evidence of recurrence, treated cervical dysplasia or treated in situ Grade 1 cervical cancer.
* Subject with unstable angina, New York Heart Association class III or IV heart failure, myocardial infarction, stroke, or deep venous thrombosis within the last 12 months; or subjects currently receiving anticoagulants.
* Subject with QT interval corrected for heart rate according to Fridericia's formula > 470 msec (females) and > 450 msec (males) during the Screening Period, confirmed by a repeat assessment.
* Subject with uncontrolled hypertension
* Subject receiving chronic treatment with more than 325 mg aspirin per day.
* Subject that requires or may require systemic immunosuppressive or immunomodulatory treatment.
* Subject who received any investigational therapy within 30 days or 5 half-lives (whichever is longer) prior to screening.
* Subject who is pregnant or breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2021-10-26 (Actual); Study Completion 2021-10-26 (Actual)

PRIMARY OUTCOMES:
Mean percentage change in serum uric acid (sUA) levels | Baseline to the end of the 4-week Dose Evaluation Period

SECONDARY OUTCOMES:
Change in mean sUA | Baseline to the end of the 4-week Dose Evaluation Period
Mean percentage change and change in mean sUA between cohorts | Baseline to the end of the 4-week Dose Evaluation Period
Percentage of patients achieving sUA of < 6.0 mg/dL (0.357 mmol/L), < 5.0 mg/dL (0.297 mmol/L), and < 4.0 mg/dL (0.238 mmol/L) | Baseline to the end of the 4-week Dose Evaluation Period
Change in mean sUA compared between BID and QD dosing | Baseline to the end of the 4-week Dose Evaluation Period

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (5):
  - Paratus - Canberra Clinic, Canberra
  - Paratus - Central Coast Clinic, Kanwal
  - Peninsula Private Hospital, Kippa-Ring
  - Emeritus Research - Melbourne, Melbourne
  - Paratus - Western Sydney Clinic, Sydney